CLINICAL TRIAL: NCT06507397
Title: Dural Puncture Epidural Anesthesia Versus Traditional Spinal Anesthesia for Rigid Cystoscopy: A Randomized Controlled Trial
Brief Title: Dural Puncture Epidural Anesthesia Versus Traditional Spinal Anesthesia for Rigid Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rabab Mohamed Mohamed Mohamed, Assistant Professor of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35621/8/22
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Dural Puncture Epidural Anesthesia; Spinal Anesthesia; Rigid Cystoscopy
MeSH Terms: interventions — Fentanyl; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Anesthesia (Active Comparator): Patients received 3-ml hyperbaric bupivacaine 0.5% and 25 mcg fentanyl (0.5-ml).
  Interventions: Drug: hyperbaric bupivacaine and fentanyl
- Dural Puncture Epidural Anesthesia (Experimental): Patients received 15-ml mixture of bupivacaine 0.25% and 50 mcg fentanyl over 5 minutes , injected in the epidural space by epidural catheter at L3-L4 interspace, a dural puncture was created by the spinal needle. Braun's Espocan® combined spinal epidural kit before insertion of epidural catheter (needle-through-needle technique) but intrathecal medication administration was withheld.
  Interventions: Drug: plain bupivacaine and fentanyl

INTERVENTIONS:
Drug: hyperbaric bupivacaine and fentanyl — Patients received 3ml hyperbaric bupivacaine 0.5% combined with 25 microg of fentanyl.
  Other Names: Spinal Anesthesia
  Arms: Spinal Anesthesia
Drug: plain bupivacaine and fentanyl — Patients received 15 mL mixture of (0.25% plain bupivacaine and 50 µg fentanyl) over 5 minutes, injected in the epidural space by epidural catheter at L3-L4 interspace, a dural puncture was created by the spinal needle. Braun's Espocan® combined spinal epidural kit before insertion of epidural catheter (needle-through-needle technique) but intrathecal medication administration was withheld.
  Other Names: Dural Puncture Epidural Anesthesia
  Arms: Dural Puncture Epidural Anesthesia

SUMMARY:
The main objective of this study was to determine if the dural puncture epidural (DPE) anesthesia provides superior analgesia and better patient satisfaction when compared to traditional spinal anesthesia for rigid cystoscopy.

DETAILED DESCRIPTION:
Most urologic surgeries are performed in a narrow and limited space with the minimally invasive technique or cystoscope, and most patients undergoing urologic surgeries are elderly individuals with other diseases.

Cystoscopic evaluation of the lower urinary tract is a vital part of an office-based urologic practice. However, regular surveillance cystoscopy is a significant source of morbidity for patients, and therefore attempts have been made to minimize discomfort secondary to this procedure.

Spinal anesthesia is popular for endoscopic urological surgery because of early recognition of symptoms caused by overhydration, transurethral resection of prostate (TURP) syndrome and bladder perforation.

The dural puncture epidural (DPE) technique is a modification of the combined spinal epidural (CSE) technique, where a dural perforation is created from a spinal needle but intrathecal medication administration is withheld. The DPE technique has been shown to improve caudal spread of analgesia compared with epidural (EPL) technique without the side effects observed with the CSE technique.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Both sex.
* American Society of Anesthesiology (ASA) physical status I, II, III.
* Admitted for elective rigid cystoscopy.

Exclusion Criteria:

* Refusal of patients.
* Body Mass Index (BMI) > 35.
* Patients who have history of substance abuse.
* Patients with difficult communication.
* Contraindication to neuraxial anesthesia (e.g.; infection near the site of injection, coagulopathy or bleeding disorder).
* Patients with history of allergy to local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the onset of anesthesia | Every 15 minutes till end of the surgery
  Assessment of the onset by test sensory loss at T10 by pin prick using sterile needle with blunt edge (defined as time from end of injection of bolus dose to 1st sign of sensory block at T10).
  Sensory level of the techniques which was assessed at 2 min after end of injection of the drug then every 5 min till the 30 min then every 15 min till end of the surgery.

SECONDARY OUTCOMES:
Time of onset of motor block | Till the end of the surgery
  Time of onset of motor block was assessed from end of drug injection to time of achieving Breen Modified Bromage scale (BMBS) grade 1) in the lower extremities was assessed by using a BMBS: Grade 1 as complete motor block to Grade 6 as no motor block) and it was assessed at 2 min then every 3 min after injection of the drug till 30 min then every 15 min till the end of the surgery.
Incidence of side effects | 24 hours postoperatively
  Incidence of side effects such as (hypotension and bradycardia) were recorded.
Number of patients required rescue analgesia | 24 hours postoperatively
  Number of patients required rescue analgesia was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.